CLINICAL TRIAL: NCT05241587
Title: Evaluation of the Effect of Xylitol Gum on Thirst, Dry Mouth and Nausea in Patients Undergoing Haemodialysis
Brief Title: Chewing Gum in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem Sarımehmet (Other)
Responsible Party: Sponsor-Investigator, Didem Sarımehmet, Lecturer, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nurse_haemo01
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Mouth Dryness; Nausea; Hemodialysis Complication; Nurse's Role; Thirst
MeSH Terms: conditions — Xerostomia; Nausea

STUDY DESIGN:
Intervention Model Description: This was a prospective, non-randomized experimental study involving a control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The chewing gum group (Experimental): Gum group patients consisted of patients who chewed "Xylitol Granule Filled Dragee Sugar Free Gum/Xylitol Gum/First X-Fresh". It is reported that the use of xylitol five times a day (not less than three times) is appropriate and effective (Xylitol, 2020; Xylitol, 2006; Llop, et al., 2010). Therefore, this group of patients was allowed to chew xylitol gum for 10 minutes, five times a day for six weeks.
  Interventions: Other: Gum Group:
- The mouth spray group (Experimental): The patients in the mouth spray group included those who had been using Oral Spray/Act Dry Mouth Spray regularly as two puffs three times a day at the request of the physician for the last two weeks. This group of patients continued to use the mouth spray at the physician's request.
  Interventions: Other: Mouth Spray Group:

INTERVENTIONS:
Other: Gum Group: — Gum Group:
  Gum group patients consisted of patients who chewed "Xylitol Granule Filled Dragee Sugar Free Gum/Xylitol Gum/First X-Fresh". It is reported that the use of xylitol five times a day (not less than three times) is appropriate and effective (Xylitol, 2020; Xylitol, 2006; Llop, et al., 2010).
  Arms: The chewing gum group
Other: Mouth Spray Group: — Mouth Spray Group:
  The patients in the mouth spray group included those who had been using Oral Spray/Act Dry Mouth Spray regularly as two puffs three times a day at the request of the physician for the last two weeks. This group of patients continued to use the mouth spray at the physician's request.
  Arms: The mouth spray group

SUMMARY:
This study was conducted to evaluate the effect of chewing xylitol gum on thirst, dry mouth and nausea in patients undergoing haemodialysis.Patients undergoing haemodialysis often experience thirst, dry mouth and nausea.This was a prospective, non-randomized experimental study involving a control group. The study was carried out with patients undergoing haemodialysis in a private dialysis centre in the northeast of Turkey between July and December 2018. It was completed with a total of 75 patients assigned to the gum group (n=25), mouth spray group (n=25), and control group (n=25).The patients in the gum group chewed xylitol gum for 10 minutes, five times a day for six weeks. Patients in the mouth spray group used two puffs of mouth spray three times a day. No intervention was made in the control group. Data were collected with the Patient Information Form, Charlson Comorbidity Index, Visual Analogue Scale, Rhodes Index of Nausea, Vomiting and Retching, graduated tube, and pH meter. Data were evaluated with Mann-Whitney U, Pearson Chi-square, Kruskal Wallis and Friedman tests. TREND checklist for non-randomised controlled trials was followed.

DETAILED DESCRIPTION:
Haemodialysis is the most preferred method in the treatment of kidney failure in the world and in Turkey. According to the 2019 reports of the United States renal data system, haemodialysis is applied to 86.9% of the chronic kidney patients. In Turkey, this rate was 74.8% as of the end of 2018, according to the data reports of the Turkish Society of Nephrology. Patients undergoing haemodialysis have to cope with the adverse effects of the chronic disease as well as complications that develop due to treatment. Causes such as drugs used in haemodialysis treatment, fluid restriction, high ultrafiltration, weight gain between two haemodialysis sessions, dialysis imbalance syndrome and deterioration of oral pH, cause fluid-electrolyte imbalances, hypotension, pain, muscle cramps, thirst, dry mouth and leads of bothersome symptoms such as nausea. These may increase morbidity and mortality by causing premature termination of haemodialysis treatment or dialysis failure. Patients undergoing haemodialysis should be able to alleviate thirst, dry mouth and nausea with a method that does not disrupt fluid restriction. The combination of the salivary gland stimulant effect of the refreshing xylitol alone together with the mechanical effect of chewing gum has the effect of reducing thirst and dry mouth. Effective in reducing thirst, dry mouth and nausea in patients undergoing haemodialysis and a method that nurses can choose independently, xylitol gum can be easily used as a safe method and increases intraoral pH, prevents oral mucositis, facilitates periodontal healing and contributes to an effective treatment process. Thirst, dry mouth and nausea are quite common bothersome symptoms in patients undergoing haemodialysis. Thirst is a symptom associated with the desire to drink water due to insufficient body fluids and is one of the body's defence mechanisms. The inability of the saliva secreted to maintain the moistness of the oral mucosa is defined as "thirst". Thirst is controlled centrally and perceived peripherally as the feeling of dry mouth. According to Bots et al., 47.8% of patients on haemodialysis were thirsty during the day, 41.6% felt thirsty before dialysis, 24.7% during dialysis and 29.9% after dialysis. Dry mouth is a symptom that results from excessive reduction in the amount of saliva or problems with secretion, usually due to under-functioning of the salivary glands. When the amount of saliva decreases below 0.1 mL/min when evaluated together with clinical symptoms, it is defined as "dry mouth (xerostomia)". Bots et al. determined that 76.4% of the patients on haemodialysis treatment experienced dry mouth, while this figure was 56.2% according to Akgöz and Arslan. Thirst and dry mouth in patients on haemodialysis causes several clinical symptoms such as the sensations of sticky or burning tongue, need to drink liquid, difficulty swallowing solid food, stomatitis, increased dental caries, dysarthria and night sleep interruptions. Nausea is the conscious recognition of the excitation of a part of the vomiting centre or a closely related area and subjective feeling of the need to vomit. Increased urea concentration in the saliva of the patients and worsening of oral pH and exposure of the oral cavity to pathogens increase the risk of developing infection, disrupt the integrity of the mucous membrane and intensify the feeling of nausea Of the patients on haemodialysis treatment, 21-54% according to Almutary and 41% according to Akgöz and Arslan experienced nausea. Uncontrollable nausea can cause undesirable symptoms such as fluid-electrolyte imbalance, dehydration, vomiting, anorexia and weight loss, and also reduce the absorption and excretion of drugs used in the treatment. Based on the previous studies in the literature, xylitol gum, used generally as an auxiliary product in providing oral hygiene and preventing dental plaques and caries, has proven effects such as increasing saliva pH, protecting salivary proteins, reducing mouth and nasopharyngeal infections and protecting mucous membrane integrity. With its refreshing and pleasant taste, xylitol gum is also recommended as a natural, economical, easily accessible and safe product for reducing thirst, dry mouth and nausea in patients undergoing haemodialysis. However, studies evaluating the effect of xylitol gum on thirst and dry mouth in patients undergoing haemodialysis are limited in both the national and international literature. In addition, studies conducted with different sample groups and different methods (patients who underwent laparoscopic breast surgery, colonoscopy preparation, gynaecological operations) concluded that chewing gum reduces nausea but no study evaluating the effect of xylitol gum on nausea in patients undergoing haemodialysis could be found.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older,
* being able to speak and understand Turkish,
* being oriented to person, place and time,
* receiving haemodialysis treatment for at least three months,
* experiencing dry mouth, thirst and nausea,
* not having any chewing difficulties,
* not having any dental prosthesis for the gum group,
* using mouth spray for the last two weeks at the request of the physician for the mouth spray group.

Exclusion Criteria:

* exclusion criteria included having a mental,
* hearing and speech impediment,
* being diagnosed with a psychiatric disease,
* using antiemetic drugs, being diagnosed with Sjögren's syndrome,
* receiving radiotherapy or chemotherapy,
* having a salivary gland infection,
* previous salivary gland surgery,
* sucking on ice cubes, chewing mint/lemon peels, and using mouthwash.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Effect of chewing xylitol gum on thirst | 6 weeks
  Thirst were evaluated with "Visual Analog Score". VAS is a 10 cm or 100 mm long measuring instrument on a horizontal line with two different ends. The left end of the line is marked as "no" and the right end as "worst".
Effect of chewing xylitol gum on dry mouth | 6 weeks
  Dry Mouth were evaluated with "Visual Analog Score". VAS is a 10 cm or 100 mm long measuring instrument on a horizontal line with two different ends. The left end of the line is marked as "no" and the right end as "worst".

SECONDARY OUTCOMES:
Effect of Xylitol Gum on nausea. | 6 weeks
  Xylitol Gum on nausea in patients undergoing haemodialysis. Nausea was evaluated with Rhodes Nausea, Vomiting and Retching Index. The highest possible value in the index is 32, which indicates the most severe symptom for the patient.
Effect of Xylitol Gum on salivary flow rate. | 6 weeks
  Xylitol Gum on salivary flow rate in patients undergoing haemodialysis. Salivary flow rate with Saliva Flow Rate Measurement Tool (Graded Tube).Saliva flow >0.25 mL/min was considered "normal"; 0.1-0.25 mL/min "low"; <0.1 mL/min "hyposalivation"
Effect of Xylitol Gum on oral pH. | 6 weeks
  Xylitol Gum on oral pH in patients undergoing haemodialysis. Salivary pH with Oral Environment pH Measurement Tool (pH Meter). When the pH meter electrode is immersed in saliva, the pH value of the saliva is determined by the pH value on the screen. "0-6 pH" appearing on the pH meter screen is considered acidic, "7 pH" neutral, and "8-14 pH" alkaline"

CONTACTS AND LOCATIONS:
Overall Officials: Didem Sarımehmet, PhD, Principal Investigator — Karadeniz Techinical University; Sevilay Hintistan, PhD, Principal Investigator — Karadeniz Techinical University
Locations (1):
- Karadeniz Techinical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almutary H, Bonner A, Douglas C. Symptom burden in chronic kidney disease: a review of recent literature. J Ren Care. 2013 Sep;39(3):140-50. doi: 10.1111/j.1755-6686.2013.12022.x. Epub 2013 Jul 4. PMID 23826803
- [Result] Akgöz N, Arslan S (2017). Examination of Symptoms in Patients Who are on Hemodialysis Treatment. Journal of Nephrology Nursing, 12(1): 20-28.